CLINICAL TRIAL: NCT03045068
Title: Platelet Transfusion During Neonatal Open Heart Surgery
Acronym: CPB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Nischal Krishamurthy Gautam, Associate Professor of Anesthesiology, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HSC-MS-16-1034
Record Dates: First submitted 2017-02-02; First posted 2017-02-07 (Estimated); Results first posted 2023-03-08 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Cardiac Disease; Cardiac Surgery; Cardiopulmonary Bypass; Platelet Transfusion; Arrythmia, Cardiac; Mortality
MeSH Terms: conditions — Heart Diseases; Arrhythmias, Cardiac | interventions — Platelet Transfusion; Platelet Count; Factor IX

STUDY DESIGN:
Intervention Model Description: Prospective Randomized trial in neonates comparing platelet apheresis transfusion prior to termination of CPB versus standard transfusion of platelet apheresis after modified ultrafiltration and protamine administration
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study Group (Experimental): Platelet Transfusion Management
  1. Pre-Termination of CPB- Platelet Transfusion 10ml/kg to be administered to the patient via central venous access when the patient has been rewarmed to 35*C, (the Sano or BT shunt clip is still on in children with SV physiology)
  2. Post CPB- Platelet transfusion 10ml/kg via a central venous line is continued at a rate of 100 ml/hour till completion.
  Interventions: Biological: Platelet Transfusion; Biological: FFP and Cryoprecipitate; Biological: PRBC and cell saver Transfusion; Biological: Factor Concentrate (Bebulin)
- Control Group (Active Comparator): Platelet Transfusion Management
  1. Pre-Termination of CPB- No intervention
  2. Post CPB- Platelet transfusion 20ml/kg via a central venous line is continued at a rate of 100 ml/hour till completion.
  Interventions: Biological: Platelet Transfusion; Biological: FFP and Cryoprecipitate; Biological: PRBC and cell saver Transfusion; Biological: Factor Concentrate (Bebulin)

INTERVENTIONS:
Biological: Platelet Transfusion — Post CPB- Platelet transfusion 20ml/kg via a central venous line is continued at a rate of 100 ml/hour till completion.
  1. Initial transfusion to occur proximal to the hemofilter on the MUF circuit for as long as MUF lasts
  2. Subsequent platelet transfusion continued till completion via central venous access to the patient
  Other Names: Platelet
Biological: FFP and Cryoprecipitate — 1. 1 unit of cryoprecipitate administered during MUF and or after MUF as needed
  2. FFP transfusion 10ml/kg during MUF and or after MUF as needed
  Other Names: FFP
Biological: PRBC and cell saver Transfusion — 1. Transfuse for target Hematocrit > 40 in neonates with SV physiology; Transfuse for Hematocrit> 33 for 2-Ventricle physiology
  Other Names: PRBC
Biological: Factor Concentrate (Bebulin) — 1. Based on clinical bleeding and achievement of hemostasis
  Other Names: Bebulin

SUMMARY:
Hypothesis:

Dilutional thrombocytopenia after cardiopulmonary bypass (CPB) is universal and administration of donor apheresis platelets just prior to termination of bypass will assist in early correction of coagulopathy, early hemostasis and lesser donor exposure of blood products after cardiac surgery.

Background:

What is the Problem? - Bleeding, Transfusion and Outcomes

1. Excessive bleeding after neonatal cardiac surgery has been independently associated with increased adverse events, morbidity and mortality.1,2 Bleeding after neonatal open-heart surgery has multiple etiologies such as immaturity of the building blocks of coagulation, effects of deep hypothermia, longer CPB times, altered flow states and dilutional state induced by being on CPB leading to low platelet count, low platelet function, low fibrinogen levels, altered fibrinogen polymerization, complement activation, etc.2,3 The strongest predictor of transfusion after cardiopulmonary bypass in children was deemed to be the CPB circuit volume and the effect of hemodilution.4
2. The dilutional coagulopathy after neonatal CPB requires intense damage control resuscitation with massive transfusion of platelets, packed red blood cells (PRBC), cryoprecipitate, fresh frozen plasma (FFP) and supplemental factor concentrates. In a previous study at this institution (IRB# HSC-MS-13-0647), we have shown that in neonates undergoing open-heart surgery there was a significant drop in platelet counts after bypass (71% change, baseline= 268 ± 90, Post CPB= 76 ± 27, 109/L). Associated with this drop , the average intraoperative transfusion load in neonates undergoing cardiac surgery with CPB at our institution constitutes of PRBC= 63± 43 ml/kg, FFP=51± 21 ml/kg, cryoprecipitate =12+6 ml/kg, platelets = 28 +16 ml/kg and cell-saver =27± 10 ml/kg. In addition 72% of these patients were exposed to a 3-factor prothrombin complex concentrate (Bebulin®). Although this "throw the kitchen sink" approach is effective in achieving hemostasis, it comes with significant effects on post CPB hemodynamics, constantly changing hematocrit, variable blood volume with inability to achieve steady state inotropic state affecting cardiac output, oxygen delivery and adding to pulmonary hypertension.

Overall, having higher platelet counts at the time of weaning from cardiopulmonary bypass has distinct advantages of reducing transfusions and improving outcomes.

DETAILED DESCRIPTION:
What do we do at our institution? The vast majority of centers including ours continue to utilize a regimen for neonatal CPB prime that constitutes of PRBCs ( 20-30 ml/kg) added to achieve a hematocrit > 25 on CPB and FFP (20-30 ml/kg) to assist the lower antithrombin levels, improve heparin efficiency and improved suppression of the thrombin generation on CPB. Platelets are not added in the CPB prime at our institution. This regimen of avoiding donor apheresis platelets transfusion during early CPB is because of the known effects of CPB on native platelets resulting in decreases in count from hemodilution and mechanical damage. Donor apheresis platelets administered as an initial constituent of CPB prime also carry the risk of platelet activation during hypothermia and CPB with potential activation of the coagulation cascade. Fresh whole blood is also not used secondary to the difficulty and logistics pertaining to availability fresh whole blood makes this approach unattractive.

What is the advantage of adding platelet apheresis just prior to separation from CPB? We know that native platelets are significantly reduced in count and function with increasing duration of CPB and function diminishes independently of platelet count with hypothermia.11 The advantages of adding donor apheresis platelets just prior to separating from CPB are that the donor platelets don't get spalliated and deformed by the roller pumps for long durations, they are not subjected to the intense cooling and rewarming process and spared of the early reperfusion injury/inflammation. Furthermore, addition of 10 ml/kg of platelets would raise the platelet counts by at least 50% based on a previous study at this institution (IRB# HSC-MS-13-0647; post-CPB platelet transfusion of 28 ± 16 ml/kg resulted in elevation of platelet counts from 76 ± 27 to 223 ± 60 (109/L).

Effect of modified ultrafiltration (MUF): MUF is routinely performed immediately on termination of CPB and prior to protamine administration. During this stage, after successful weaning from CPB, 10-15% of the cardiac output from the arterial cannula along with residual volume from the venous reservoir of the CPB pump is pumped through a hemofilter placed under vacuum to allow rapid hemofiltration with the effluent returned via a single atrial venous cannula to the patient. This 15-minute rapid hemofiltration allows for removal of excess water, improvement in hematocrit with improved oxygen delivery, faster achievement of steady state inotrope levels with improved hemodynamics and removal of inflammatory mediators.12-14 While MUF improves hematocrit, it does not increase platelet count significantly, MUF has no effect on native platelet function.3 The biggest advantage of transfusion of apheresis platelets prior to termination of bypass versus standard practice of their transfusion after protamine is that the transfused fluid load of 10-15 ml/kg of platelets volume that would have diluted the red cell fraction (hematocrit) and impacted oxygen delivery and pulmonary dysfunction would now take the full benefit of modified ultrafiltration with excess fluid removal even prior to protamine administration with overall improved hemodynamics.

Institutional Blood transfusion Management for Neonatal CPB For the CPB prime: PRBCs (50ml/kg) are added to allow for a hematocrit >30 for the estimated blood volumes. FFP is added to the pump prime for all patients weighing less than 5 kilograms and in those who demonstrate heparin resistance on initial heparin dose response assays. Heparin is added in the CPB prime. Other constituents of the CPB prime are epsilon aminocaproic acid (50 mg/kg), cefazolin (30 mg/kg) and methylprednisolone.

Post CPB: Current practice in neonates is to administer a combination of cryoprecipitate, platelet and PRBC in a 1:1:1 ratio till hemostasis is achieved. 3PCC factor administration is based on diffuse clinical bleeding suggestive of coagulopathy that persists despite one round of cryoprecipitate and platelet transfusion.

Study Method:

Prospective Randomized trial in neonates comparing platelet apheresis transfusion prior to termination of CPB versus standard transfusion of platelet apheresis after modified ultrafiltration and protamine administration. Primary outcomes and secondary outcomes are detailed below.

Study Group Platelet Transfusion Management

1. Pre-Termination of CPB- Platelet Transfusion 10ml/kg to be administered to the patient via central venous access when the patient has been rewarmed to 35*C, (the Sano or BT shunt clip is still on in children with SV physiology)
2. Post CPB- Platelet transfusion 10ml/kg via a central venous line is continued at a rate of 100 ml/hour till completion.

FFP and Cryoprecipitate:

1. 1 unit of cryoprecipitate administered during MUF and or after MUF as needed
2. FFP transfusion 10ml/kg during MUF and or after MUF as needed

PRBC and cell saver Transfusion:

1. Transfuse for target Hematocrit > 40 in neonates with SV physiology; Transfuse for Hematocrit> 33 for 2-Ventricle physiology

3- Factor Concentrate (Bebulin):

1. Based on clinical bleeding and achievement of hemostasis

Control Group Platelet Transfusion Management 1. Pre-Termination of CPB- No intervention 2. Post CPB- Platelet transfusion 20ml/kg via a central venous line is continued at a rate of 100 ml/hour till completion.

1. Initial transfusion to occur proximal to the hemofilter on the MUF circuit for as long as MUF lasts
2. Subsequent platelet transfusion continued till completion via central venous access to the patient

   FFP and Cryoprecipitate:
   1. 1 unit of cryoprecipitate administered during MUF and or after MUF as needed
   2. FFP transfusion 10ml/kg during MUF and or after MUF as needed

   PRBC and cell saver Transfusion:

   1. Transfuse for target Hematocrit > 40 in neonates with SV physiology; Transfuse for Hematocrit> 33 for 2-Ventricle physiology

   3 Factor Concentrate (Bebulin):
   1. Based on clinical bleeding and achievement of hemostasis

      Objectives

      a) Volume of Blood Transfusion (PRBC, FFP, Cryo, Platelets) Number of Donor Exposures (PRBC, FFP, Cryo, Platelets) from termination of CPB to first 24 hours post op b) Number of exposures of 4-PCC and Factor 7 c) Time from termination of CPB to Chest Approximation
      1. Chest tube output first 24 hours
      2. Inotropic support at time of chest approximation and at 24 hours postop
      3. Length of mechanical ventilation
      4. 30 day mortality
      5. Mediastinal exploration
      6. Delayed sternal closure
      7. Perioperative cardiac arrest first 72 hours
      8. Arrhythmia

      Sample size- Based on pilot data we have collected in the standard procedure group, the mean and standard deviation (SD) of total blood product intake during first 24 hours is 125.3+/- 71.1 (ml/kg). To detect a 1*SD unit reduction on the total blood intake, we need 17 patients per group with 80% power at 0.05 significance level. To account for 20% drop out rate, we need 22 patients per group, i.e. 44 patients in total.

      Inclusion Criteria- All neonates and infants less than 3 months of age under 4 kilograms undergoing open heart surgery and cardiopulmonary bypass.

      Exclusion Criteria-1) Redo open heart surgery 2) Bleeding Disorders - such as von Willebrand Disease, Hemophilia

      Screening and Recruitment:

      The list of newborns to be operated will be obtained daily from the operating room log.

      Care4 records and OR Tracking will be used to screen for patients Initials of Patients, Date of Brith, Date of Surgery and MRN will be collected. The Research Team ( PI and Co-PI) will make contact with the family member while obtaining the surgical and or the anesthesia consent.

      Data Collected ( routine Standard operating procedure data)

      Patient Demographics:

      MRN, Gestational age, Age at operation, weight at birth, weight at operation, primary Diagnosis, Other diagnosis,

      Operative Data:

      CPB time, Aortic Cross Clamp time, Deep Hypothermic Circulatory Arrest time, Antegrade Cerebral perfusion time, Case duration.

      Pump Prime Constituents:

      Inotrope score: at chest approximation {dopamine + dobutamine + (epinephrine*100) + (milrinone*10) 15 Procedure performed. Complications All Laboratory values performed from baseline to 24 hours postoperative

      a) Baseline- CBC with Platelets, Fibrinogen, TEG b) Rewarming, prior to termination at core temperature of 35*C- CBC with platelets, Fibrinogen, TEG c) Arrival to PICU- CBC with platelets, fibrinogen, TEG d) 24 hours post op- CBC with platelets, fibrinogen, TEG All Blood products administered with age of the blood product at time of administration (<5 days, > 5days) Post operative Length of Intubation STS reportable complications Mortality Cumulative fluid balance first 72 hours.

      Outcome Variables:

      d) Number of Donor Exposures (PRBC, FFP, Cryo, Platelets) from termination of CPB to first 24 hours post op e) Number of exposures of 4-PCC and Factor 7 f) Time from termination of CPB to Chest Approximation i) Chest tube output first 24 hours j) Inotropic support at time of chest approximation and at 24 hours postop k) Length of mechanical ventilation l) 30 day mortality m) Mediastinal exploration n) Delayed sternal closure o) Perioperative cardiac arrest first 72 hours p) Arrhythmia

      Study Risks:

      There are no perceivable risks from exposure to platelets since the patients will be exposed to platelet transfusion after protamine administration. Only the timing of administration is being changed in the study group.

      Informed Consent:

      A written informed consent will be obtained. If informed consent is not obtainable or refused, patients will be randomized to control arm.

ELIGIBILITY:
Inclusion Criteria:

All neonates and infants less than 3 months of age under 4 kilograms undergoing open heart surgery and cardiopulmonary bypass

Exclusion Criteria:

1. Redo open heart surgery
2. Bleeding Disorders - such as von Willebrand Disease, Hemophilia

Ages: 1 Day to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2017-04-11 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nischal K Gautam, MD, Principal Investigator — The University of Texas Health Science at Houston
Locations (1):
- Memorial Hermann Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Group: Platelet Transfusion Management
  1. Pre-Termination of CPB- Platelet Transfusion 10ml/kg to be administered to the patient via central venous access when the patient has been rewarmed to 35*C, (the Sano or BT shunt clip is still on in children with SV physiology)
  2. Post CPB- Platelet transfusion 10ml/kg via a central venous line is continued at a rate of 100 ml/hour till completion.
  Platelet Transfusion: Post CPB- Platelet transfusion 20ml/kg via a central venous line is continued at a rate of 100 ml/hour till completion.
  1. Initial transfusion to occur proximal to the hemofilter on the MUF circuit for as long as MUF lasts
  2. Subsequent platelet transfusion continued till completion via central venous access to the patient
  FFP and Cryoprecipitate: 1. 1 unit of cryoprecipitate administered during MUF and or after MUF as needed 2. FFP transfusion 10ml/kg during MUF and or after MUF as needed
  PRBC and cell saver Transfusion: 1. Transfuse for target Hematocrit > 40 in neonates with SV physiology; Transfuse for Hematocrit> 33 for 2-Ventricle physiology
  Factor Concentrate (Bebulin): 1. Based on clinical bleeding and achievement of hemostasis
- Control Group: Platelet Transfusion Management
  1. Pre-Termination of CPB- No intervention
  2. Post CPB- Platelet transfusion 20ml/kg via a central venous line is continued at a rate of 100 ml/hour till completion.
  Platelet Transfusion: Post CPB- Platelet transfusion 20ml/kg via a central venous line is continued at a rate of 100 ml/hour till completion.
  1. Initial transfusion to occur proximal to the hemofilter on the MUF circuit for as long as MUF lasts
  2. Subsequent platelet transfusion continued till completion via central venous access to the patient
  FFP and Cryoprecipitate: 1. 1 unit of cryoprecipitate administered during MUF and or after MUF as needed 2. FFP transfusion 10ml/kg during MUF and or after MUF as needed
  PRBC and cell saver Transfusion: 1. Transfuse for target Hematocrit > 40 in neonates with SV physiology; Transfuse for Hematocrit> 33 for 2-Ventricle physiology
  Factor Concentrate (Bebulin): 1. Based on clinical bleeding and achievement of hemostasis
Period: Overall Study
Arm/Group | Study Group | Control Group
Started | 23 | 23
Received Intervention | 23 | 23
Completed | 21 | 21
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Study Group | Control Group | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Continuous [Mean (Standard Deviation); unit: Days] | 8.1 (3) | 9.3 (7) | 8.7 (5)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: This data was not collected.
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 21 | 21 | 42
Weight [Mean (Standard Deviation); unit: kilograms]
  Weight at birth | 3.1 (0.4) | 3.0 (0.5) | 3.05 (0.45)
  Weight at surgery | 3.1 (0.4) | 3.1 (0.5) | 3.1 (0.45)
Number of participants with presence of genetic syndrome [Number; unit: participants] | 4 | 4 | 8
Number of participants with baseline oxygen saturation < 90% [Count of Participants; unit: Participants] | 10 | 11 | 21
The Society of Thoracic Surgeons-European Association for Cardio-Thoracic Surgery (STAT) score [Count of Participants; unit: Participants] — The STAT score is a tool designed to analyze the risk for mortality associated with different types of congenital heart surgery procedures. Categories range from Category 1 to Category 5--procedures associated with lowest mortality rates are in Category 1, and procedures associated with highest mortality rates are in Category 5.
  Participants
    Number of participants with STAT score of 2 | 1 | 0 | 1
    Number of participants with STAT score of 3 | 4 | 4 | 8
    Number of participants with STAT score of 4 | 11 | 9 | 20
    Number of participants with STAT score of 5 | 5 | 8 | 13
Platelet count, pre-cardiopulmonary bypass (CPB) [Mean (Standard Deviation); unit: K/cmm] | 288 (87) | 246 (106) | 267 (96.5)
Fibrinogen, pre-cardiopulmonary bypass (CPB) [Mean (Standard Deviation); unit: milligram per deciliter (mg/dL)] | 267 (75) | 248 (50) | 257.5 (62.5)
Maximal amplitude on kaolin-heparinase thromboelastography (MA [TEG]), pre-CPB [Mean (Standard Deviation); unit: millimeter (mm)] — The TEG assay assesses clot properties, and the the maximal amplitude (MA) as assessed by TEG reflects platelet contribution to clot strength. Low MA values correspond with states of platelet dysfunction or hypofibrinogenemia.
  millimeter (mm) | 65 (7) | 63 (7) | 64 (7)

OUTCOME MEASURES:

1. Primary Outcome: Amount of Blood Products Transfused
Description: All Blood products administered (PRBC, FFP, Cryo, Platelets) from termination of CPB to first 24 hours post op
Time Frame: 0-72 hours
Measure: Mean (Standard Deviation); unit: milliliter per kilogram (mL/kg)
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 21 | 21
milliliter per kilogram (mL/kg) | 58 (29) | 103 (80)

2. Secondary Outcome: Number of Exposures of 4-PCC and Factor 7
Description: Number of exposures of 4-PCC and Factor 7
Time Frame: 0-72 hours
Measure: Number; unit: exposures
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 21 | 21
exposures | 5 | 6

3. Secondary Outcome: Time From End of CPB to Sternal Closure (Chest Approximation)
Description: This outcome reports the time from the end of the cardiopulmonary bypass (CPB) procedure to the time the sternum is closed.
Time Frame: 0-72 hours
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 21 | 21
days | 1.48 (0.98) | 1.95 (1.20)

4. Secondary Outcome: Chest Tube Output
Description: A chest tube is a flexible tube used to drain fluid or air from the chest, and the amount removed over 24 hours will be reported.
Time Frame: 0-24 hours
Measure: Mean (Standard Deviation); unit: milliliter per kilogram (mL/kg)
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 21 | 21
milliliter per kilogram (mL/kg) | 20 (11) | 23 (18)

5. Secondary Outcome: Inotropic Support at the Time of Entry to the Pediatric Intensive Care Unit (PICU) as Indicated by Inotrope Score
Description: The inotrope score equals [dopamine dose (mg/kg/min) + dobutamine dose (mg/kg/min) + epinephrine dose (mg/kg/min) X100 + milrinone (mg/kg/min) x 10]. A higher score indicates that the patient is in more critical condition and requires a greater level of treatment. The score ranges from 0 to about 90.
Time Frame: At the time of entry to the pediatric intensive care unit (PICU)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 21 | 21
score on a scale | 7.1 (3.7) | 5.6 (2.9)

6. Secondary Outcome: Length of Mechanical Ventilation
Time Frame: from start of mechanical ventilation to end of mechanical ventilation (about 4-8 days)
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 21 | 21
days | 4.1 (1.8) | 8 (6.7)

7. Secondary Outcome: Number of Participants With Mortality at 30 Days
Description: 30 day mortality
Time Frame: 0-30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 21 | 21
Participants | 0 | 0

8. Secondary Outcome: Number of Participants With Cardiopulmonary Resuscitation (CPR) Events
Description: Perioperative cardiac arrest first 72 hours
Time Frame: 0-72 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 21 | 21
Participants | 0 | 4

9. Secondary Outcome: Number of Participants With Arrhythmia
Description: Arrhythmia
Time Frame: 0-72 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 21 | 21
Participants | 3 | 6

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Study Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21 | 4/21
Other Adverse Events (participants affected / at risk) | 3/21 | 6/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Group (N=21) | Control Group (N=21)
Cardiopulmonary Resuscitation (CPR) Event (General disorders) | 0 (0) | 4 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Group (N=21) | Control Group (N=21)
Arrhythmia (Cardiac disorders) | 3 (3) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-04): https://cdn.clinicaltrials.gov/large-docs/68/NCT03045068/Prot_SAP_000.pdf